CLINICAL TRIAL: NCT02701816
Title: Korean Multicenter Registry of INNOVA Stent for Femoropopliteal Artery Disease: (K-INNOVA Registry)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2015-0074
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Femoropopliteal Artery Disease
Keywords: Peripheral Artery Disease; Femoropopliteal Artery; Nitinol Stent; Restenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- K-INNOVA: Patients with femoropopliteal artery disease undergoing endovascular therapy using Innova stent (Boston Scientific).
  Interventions: Device: innova stent (Boston scientific)

INTERVENTIONS:
Device: innova stent (Boston scientific)

SUMMARY:
* Prospective, single-arm, multi-center registry study
* A total of 150 subjects with femoropopliteal artery disease who meet all inclusion and exclusion criteria will be included.
* Patients will be followed clinically for 12 months after the procedure.
* Duplex ultrasound, CT or catheter-based angiography follow-up according to participating hospital's protocol will be performed at 12 months.
* Presence of stent fracture will be evaluated by plain radiography or fluoroscopy at 12 months.
* Quality of life by standardized questionnaires (at baseline & at 1 & 12 months)

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years of older
2. Symptomatic peripheral artery disease:

   * Moderate or severe claudication (Rutherford category 2 or 3)
   * Critical limb ischemia (Rutherford category 4-5)
3. Femoropopliteal artery lesions with stenosis > 50%
4. ABI < 0.9
5. Patients with signed informed consent

Exclusion Criteria:

1. Acute critical limb ischemia
2. Severe critical limb ischemia (Rutherford category 6)
3. Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, cilostazol, or contrast agents
4. In-stent restenosis lesions (Restenosis lesions without previously implanted stents are eligible to the enrollment)
5. Bypass graft lesions
6. Age > 85 years
7. Severe hepatic dysfunction (> 3 times normal reference values)
8. Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
9. LVEF < 40% or clinically overt congestive heart failure
10. Pregnant women or women with potential childbearing
11. Life expectancy <1 year due to comorbidity
12. Untreated proximal inflow disease of the ipsilateral iliac arteries (more than 50% stenosis or occlusion)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Femoropopliteal artery disease
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 12 months after the index procedure
  Absence of restenosis >50%

SECONDARY OUTCOMES:
Target lesion revascularization rate | 12 months
Stent fracture rate | 12 months
Quality of life | 12 months
  Quality of life by standardized questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No